CLINICAL TRIAL: NCT02294942
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Study to Evaluate the Effects of add-on RANCAD on Exercise Tolerance and Angina Frequency in Patients With Stable Angina Pectoris.
Brief Title: Extended-Release RANCAD in the Patients With Stable Angina Pectoris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TSHRN1201
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Stable Angina Pectoris
Keywords: RNTA06; RANCAD
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RANCAD 500mg (Experimental): RANCAD 1 tab (500 mg) + Placebo 1 tab, twice daily.
  Interventions: Drug: RANCAD
- RANCAD 1000mg (Experimental): RANCAD 2 tabs (500 mg), twice daily
  Interventions: Drug: RANCAD
- Placebo (Active Comparator): 2 tabs, twice daily
  Interventions: Drug: RANCAD

INTERVENTIONS:
Drug: RANCAD — Extended-Release RANCAD
  Other Names: RNTA06

SUMMARY:
A double-blind, randomized, placebo-controlled, parallel study to evaluate the effects of add-on RANCAD on exercise tolerance and angina frequency in patients with stable angina pectoris.

DETAILED DESCRIPTION:
Primary objective is to to determine the effects of add-on RANCAD on exercise treadmill test (ETT) duration at trough plasma level of RANCAD level after 12-weeks therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 20 years old
2. A minimum 3-month history of stable angina
3. Patients with diagnosis of coronary artery disease (CAD)
4. Patients present with the symptoms of stable angina after withdrawn from other antianginal drugs and given the required background therapy for at least 7 days will be qualified for entering this study and performing 1st ETT qualifying test
5. Patients developed exercise-induced ECG ischemiai during two qualifying exercise treadmill testsii. The difference between twoiii tests should be ≤ 20% of the longer test or ≤ 1 minute i. Exercise-induced ECG ischemia is defined as the new development of horizontal or down-sloping ST-segment depression of ≥1mm at 60-80ms after the J point; if patients with baseline ST depression at rest (<1mm), qualifying ST segment depression is defined as additional ST depression of at least 1 mm below the resting value ii. Exercise treadmill test (ETT) will be performed by Modified Bruce Protocol. iii. Two qualifying tests will be conducted 1 week apart, a 3rd ETT test will be performed ≤ 3 days when differences between previous two qualifying ETTs >20% of the longer test or >1 minute
6. Willing and able to provide a written informed consent

Exclusion Criteria:

1. Factors that might compromise ECG or ETT interpretation

   * Patients with resting ST-segment depression ≥ 1mm in any lead
   * Left bundle-branch block
   * Patients implanted with pacemaker
   * Patients under Digitalis therapy
2. Patients with family history of (or congenital) long QT syndrome
3. Patients with congenital heart disease
4. Patients with uncorrected valvular heart disease
5. Patients with unstable angina, or MI, or coronary revascularization procedure ≤ 2 months prior enter this study
6. Female who is pregnant/lactating or planning to be pregnant, or female of childbearing potential* who is not using medically recognized method of contraception

   *Other than those who have been surgically sterilized (defined as having undergone hysterectomy or bilateral oophorectomy or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal.
7. Patients are under any one of the following conditions:

   * New York Heart Association (NYHA) Class III or Class IV congestive heart failure (CHF)
   * QTc > 450 msec at screening
   * Active myocarditis, pericarditis, hypertrophic cardiomyopathy
   * Uncontrolled hypertension (defined as SBP > 180 mmHg) Voltage criteria for left ventricular hypertrophy in the absence of repolarization abnormalities will not be exclusion criteria
8. Use of any investigational product ≤ 4 weeks prior to screening
9. Patients with severe hepatic disease (e.g., liver cirrhosis)
10. Patients with impaired renal function (defined as serum Cr >1.5 mg/dl)
11. Patients with any condition or disease which is considered not suitable for this study by investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
ETT performing at last treatment visit (Week 12). | Week 12 (not including screening & follow-up period)
  To compare the change from baseline of ETT performing duration between add-on RANCAD and placebo at trough (12 hours after dosing) at Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Juey-Jen Hwang, M.D., Ph.D.,, Principal Investigator — National Taiwan University Hospital
Locations (6):
- Taiwan (6):
  - Far Eastern Memorial Hospital, New Taipei City, New Taipei city
  - Mackay Memorial Hospital, Taipei, Taipei City
  - Shin Kong WuHoSu Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District